CLINICAL TRIAL: NCT00538213
Title: Reactogenicity and Immunogenicity of GSK Biologicals' Influenza Vaccine GSK576389A in Elderly Adults (≥66 Years) Previously Vaccinated With the Same Candidate Vaccine. Fluarix™ Will be Used as Reference
Brief Title: Evaluation of Safety and Immunogenicity of GSK Bio's Influenza Vaccine GSK576389A After Repeated Vaccination in Elderly Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110263
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Influenza
Keywords: Influenza vaccine GSK576389A; Fluarix; Influenza infection
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (3):
- Adjuvanted influenza vaccine GSK576389A Group (Experimental): Subjects aged ≥ 66 years who previously received 1 dose of adjuvanted influenza vaccine GSK576389A in NCT00318149 and NCT00386698 studies were administered 1 dose of adjuvanted influenza vaccine GSK576389A.
  Interventions: Biological: GSK Bio's Influenza Vaccine GSK576389A
- Fluarix young Group (Active Comparator): Subjects aged 19-42 years who previously received 1 dose of Fluarix vaccine in NCT00318149 and NCT00386698 studies were administered 1 dose of Fluarix vaccine.
  Interventions: Biological: Fluarix™
- Fluarix elderly Group (Active Comparator): Subjects aged ≥ 66 years who previously received 1 dose of Fluarix vaccine in NCT00318149 and NCT00386698 studies were administered 1 dose of Fluarix vaccine.
  Interventions: Biological: Fluarix™

INTERVENTIONS:
Biological: Fluarix™ — Single dose, Intramuscular injection
  Arms: Fluarix elderly Group; Fluarix young Group
Biological: GSK Bio's Influenza Vaccine GSK576389A — Single dose, Intramuscular injection
  Arms: Adjuvanted influenza vaccine GSK576389A Group

SUMMARY:
Since influenza vaccines are administered every year because of the frequent change in their antigenic composition, the safety and immunogenicity profile of GSK Biologicals' influenza vaccine GSK576389A will be re-evaluated after repeated vaccine administration. In this study, the subjects previously enrolled in study 104887 will receive a dose with the 2007-2008 season's formulations of Fluarix or GSK576389A. Only subjects who were previously enrolled in study 104887 are eligible for participation in this study.

DETAILED DESCRIPTION:
This study is a year 2 revaccination study. First year revaccination was done in study 104887 (NCT00386698). Primary study was study 104886 (NCT00318149). This study involves 2 age groups (based on primary study):

Subjects enrolled in the ≥ 65 years age group in the primary study. Subjects enrolled in the 18-40 years age group in the primary study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously vaccinated with GlaxoSmithKline Biologicals Fluarix™ or GSK576389A investigational vaccines in the 104887 study (NCT00386698).
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female aged between 19 and 42 years or 66 years and older at the time of the vaccination.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by clinical evaluation before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days prior to vaccination, or planned use during the study period.
* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study. Planned administration of a vaccine not foreseen by the study protocol up to 21 days after vaccination.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Vaccination against influenza since January 2007 with the Northern Hemisphere 2007/2008 influenza vaccine or 2006/2007 influenza vaccine.
* History of confirmed influenza infection since the date of previous vaccination.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the administration of the study vaccine. (For corticosteroids, this will mean prednisone, or equivalent, ≥0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccine(s)
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by clinical evaluation (medical history and medical history directed physical examination) or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e. Axillary temperature <37.5°C / Oral temperature of <37.5°C).
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or planned administration during the study.
* Any medical conditions in which intramuscular injections are contraindicated.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-10-15; Primary Completion 2007-11-01 (Actual); Study Completion 2007-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110263 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Started | 55 | 40 | 38
Completed | 55 | 40 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group | Total
Number analyzed (Participants) | 55 | 40 | 38 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.2 (3.07) | 71.2 (3.47) | 27.4 (6.08) | 58.69 (20.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 16 | 55
  Male | 33 | 23 | 22 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, redness and swelling was greater than 100 millimeter i.e. >100 mm and grade 3 pain was considerable pain at rest that prevented normal everyday activities. Any was occurrence of any local symptom regardless of their intensity grade.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Number; unit: subjects
Groups:
- Adjuvanted Influenza Vaccine GSK576389A Group: Subjects aged ≥ 66 years who previously received 1 dose of adjuvanted influenza vaccine GSK576389A in NCT00318149 and NCT00386698 studies were administered 1 dose of adjuvanted influenza vaccine GSK576389A in this study.
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 55 | 40 | 38
subjects
  Any ecchymosis | 0 | 0 | 0
  Grade 3 ecchymosis | 0 | 0 | 0
  Any pain | 40 | 12 | 34
  Grade 3 pain | 0 | 0 | 0
  Any redness | 13 | 6 | 1
  Grade 3 redness | 0 | 0 | 0
  Any swelling | 6 | 4 | 0
  Grade 3 swelling | 0 | 0 | 0

2. Primary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 40 | 12 | 34
Days
  Pain (N=40; 12; 34) | 2.0 [1.0 to 5.0] | 1.5 [1.0 to 4.0] | 2.0 [1.0 to 4.0]
  Redness (N=13; 6; 1) | 3.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0]
  Swelling (N=6; 4; 0) | 3.0 [2.0 to 5.0] | 1.0 [1.0 to 3.0] | NA [NA to NA] — No subjects from this group reported any swelling

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any temperature was defined as axillary temperature ≥38.0 degree centigrade (°C), grade 3 temperature was axillary temperature ≥39.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relation to vaccination and grade 3 was defined as general symptom that prevented normal activity. Related was general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-6
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 55 | 40 | 38
subjects
  Any arthralgia | 6 | 6 | 2
  Grade 3 arthralgia | 0 | 0 | 0
  Related arthralgia | 4 | 3 | 2
  Any fatigue | 19 | 6 | 9
  Grade 3 fatigue | 0 | 0 | 0
  Related fatigue | 19 | 3 | 8
  Any headache | 13 | 5 | 8
  Grade 3 headache | 0 | 0 | 0
  Related headache | 11 | 2 | 7
  Any myalgia | 10 | 3 | 10
  Grade 3 myalgia | 0 | 0 | 1
  Related myalgia | 10 | 1 | 10
  Any nausea | 4 | 0 | 3
  Grade 3 nausea | 0 | 0 | 0
  Related nausea | 4 | 0 | 1
  Any shivering | 10 | 0 | 2
  Grade 3 shivering | 0 | 0 | 1
  Related shivering | 9 | 0 | 2
  Any temperature | 4 | 0 | 0
  Grade 3 temperature | 0 | 0 | 0
  Related temperature | 4 | 0 | 0

4. Primary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: Day 0-6
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 19 | 6 | 10
Days
  Arthralgia (N=6; 6; 2) | 2.5 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 1.5 [1.0 to 2.0]
  Fatigue (N=19; 6; 9) | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]
  Headache (N=13; 5; 8) | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0]
  Myalgia (N=10; 3; 10) | 2.0 [1.0 to 5.0] | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 3.0]
  Nausea (N=4; 0; 3) | 1.0 [1.0 to 2.0] | NA [NA to NA] — No subjects from this group reported any nausea | 1.0 [1.0 to 2.0]
  Shivering (N=10; 0; 2) | 1.0 [1.0 to 3.0] | NA [NA to NA] — No subjects from this group reported any shivering | 3.5 [1.0 to 6.0]
  Temperature (N=4; 0; 0) | 1.0 [1.0 to 1.0] | NA [NA to NA] — No subjects from this group reported any temperature | NA [NA to NA] — No subjects from this group reported any temperature

5. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was event that prevented normal activities and related was defined as unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 55 | 40 | 38
subjects
  Any AE(s) | 18 | 9 | 19
  Grade 3 AE(s) | 1 | 1 | 1
  Related AE(s) | 6 | 2 | 3

6. Primary Outcome: Number of Subjects Reporting at Least One, Grade 3 and Related Medically Significant Conditions (MSCs)
Description: MSCs were defined as AEs with a medically-attended visit i.e. prompting emergency room (ER) visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination. At least one MSC was defined as at least one MSC experienced. Grade 3 was MSC that prevented normal activities and Related was defined as MSC assessed by the investigator to be causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 55 | 40 | 38
subjects
  At least one MSC | 5 | 1 | 2
  Grade 3 MSC | 0 | 0 | 1
  Related MSC | 0 | 0 | 0

7. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade and related was event assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 55 | 40 | 38
subjects
  Any SAE(s) | 0 | 0 | 0
  Related SAE(s) | 0 | 0 | 0

8. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Days 0 and 21
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity were available at day 21.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 52 | 39 | 38
titer
  A/Solomon Islands strain at Day 0 (N=52; 39; 38) | 8.5 [6.7 to 10.8] | 6.9 [5.7 to 8.5] | 56.0 [35.2 to 89.1]
  A/Solomon Islands strain at Day 21 (N=51; 39; 38) | 91.6 [64.1 to 131.0] | 30.3 [18.7 to 49.2] | 110.0 [76.5 to 158.3]
  A/Wisconsin strain at Day 0 (N=52; 39; 38) | 141.9 [103.1 to 195.3] | 70.6 [47.4 to 105.2] | 115.1 [77.5 to 171.1]
  A/Wisconsin strain at Day 21 (N=51; 39; 38) | 384.5 [301.7 to 489.8] | 147.6 [105.9 to 205.6] | 190.1 [144.0 to 251.0]
  B/Malaysia strain at Day 0 (N=52; 39; 38) | 82.6 [64.7 to 105.6] | 59.6 [42.3 to 83.8] | 139.4 [98.5 to 197.2]
  B/Malaysia strain at Day 21 (N=51; 39; 38) | 163.2 [129.6 to 205.7] | 93.8 [68.4 to 128.8] | 210.3 [158.6 to 278.7]

9. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies
Description: Seropositivity was defined as antibody titer greater than or equal to the cut-off value i.e. ≥ 1:10. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 52 | 39 | 38
subjects
  A/Solomon Islands strain at Day 0 (N=52; 39; 38) | 19 | 12 | 33
  A/Solomon Islands strain at Day 21 (N=51; 39; 38) | 48 | 28 | 37
  A/Wisconsin strain at Day 0 (N=52; 39; 38) | 50 | 37 | 37
  A/Wisconsin strain at Day 21 (N=51; 39; 38) | 51 | 39 | 38
  B/Malaysia strain at Day 0 (N=52; 39; 38) | 52 | 38 | 37
  B/Malaysia strain at Day 21 (N=51; 39; 38) | 51 | 38 | 38

10. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies
Description: Seroconversion was defined as either a pre-vaccination titer <1:10 and a post-vaccination titer ≥1:40 or a pre-vaccination titer ≥1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 51 | 39 | 38
subjects
  A/Solomon Islands strain | 39 | 19 | 6
  A/Wisconsin strain | 18 | 6 | 4
  B/Malaysia strain | 10 | 4 | 2

11. Secondary Outcome: HI Antibody Seroconversion Factors (SCF)
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Day 21
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 51 | 39 | 38
fold increase
  A/Solomon Islands strain | 10.6 [7.4 to 15.2] | 4.4 [2.8 to 6.8] | 2.0 [1.5 to 2.5]
  A/Wisconsin strain | 2.7 [2.2 to 3.3] | 2.1 [1.7 to 2.5] | 1.7 [1.4 to 2.0]
  B/Malaysia strain | 2.0 [1.7 to 2.3] | 1.6 [1.3 to 1.9] | 1.5 [1.3 to 1.8]

12. Secondary Outcome: The Number of Subjects Seroprotected to HI Antibodies
Description: Seroprotection was defined as serum HI titer ≥1:40 that usually is accepted as indicating protection. The vaccine strains included A/Solomon Islands, A/Wisconsin and B/Malaysia antigens.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Number; unit: subjects
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 52 | 39 | 38
subjects
  A/Solomon Islands strain at Day 0 (52; 39; 38) | 6 | 1 | 25
  A/Solomon Islands strain at Day 21 (51; 39; 38) | 42 | 21 | 32
  A/Wisconsin strain at Day 0 (N= 52; 39; 38) | 49 | 31 | 33
  A/Wisconsin strain at Day 21 (N= 51; 39; 38) | 50 | 35 | 37
  B/Malaysia strain at Day 0 (N=52; 39; 38) | 47 | 31 | 35
  B/Malaysia strain at Day 21 (N=51; 39; 38) | 51 | 37 | 37

13. Secondary Outcome: The Geometric Mean (GM) Number of CD4 T-cells Per Million CD4+ T-cells for Each Vaccine Strain and for Pooled Vaccine Strains Producing at Least Two Different Immune Markers or Producing Each of the Immune Markers Plus Another Immune Marker
Description: The vaccine strains included A/Solomon Islands, A/Wisconsin, B/Malaysia and Pool FLU antigens and the markers assessed were Cluster of Differentiation 4-All doubles i.e. CD4-All doubles, CD40 Ligand (CD40L), interferon-gamma (IFN-γ), interleukin-2 (IL-2) and tumor necrosis factor alpha (TNF-α).
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: CD4 cells/10^6 CD4+ cells
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 44 | 36 | 36
CD4 cells/10^6 CD4+ cells
  A/Solomon Islands[CD4-All doubles] D0(N=44;36;36) | 289.37 (316.11) | 180.39 (228.07) | 331.14 (494.08)
  A/Solomon Islands[CD4-All doubles] D21(N=44;36;35) | 700.62 (634.14) | 337.23 (500.65) | 258.27 (637.94)
  A/Wisconsin[CD4-All doubles] D0 (N=44;36;36) | 603.80 (540.62) | 489.94 (426.96) | 905.24 (750.96)
  A/Wisconsin[CD4-All doubles] D21 (N=44;36;35) | 1020.35 (830.08) | 776.74 (654.62) | 868.45 (946.28)
  B/Malaysia[CD4-All doubles] D0 (N=44;35;36) | 448.88 (497.51) | 381.99 (341.08) | 566.22 (581.71)
  B/Malaysia[CD4-All doubles] D21 (N=44;36;35) | 925.46 (607.25) | 681.59 (593.45) | 786.37 (723.64)
  Pool FLU[CD4-All doubles] D0 (N=44;36;36) | 1054.11 (945.41) | 983.41 (598.15) | 1693.14 (1045.17)
  Pool FLU[CD4-All doubles] D21 (N=44;36;35) | 2115.03 (1368.50) | 1509.46 (1159.17) | 1998.24 (1287.85)
  A/Solomon Islands[CD4-CD40L] D0 (N=44;36;36) | 270.70 (307.98) | 165.45 (211.89) | 309.92 (437.51)
  A/Solomon Islands[CD4-CD40L] D21(N=44;36;35) | 642.40 (596.29) | 302.95 (473.99) | 236.63 (553.12)
  A/Wisconsin[CD4-CD40L] D0 (N=44;36;36) | 549.05 (509.04) | 447.08 (404.96) | 851.31 (663.11)
  A/Wisconsin[CD4-CD40L] D21 (N=44;36;35) | 930.92 (790.99) | 709.71 (622.14) | 726.97 (809.91)
  B/Malaysia[CD4-CD40L] D0 (N=44;35;36) | 429.49 (476.96) | 332.83 (337.05) | 595.14 (562.39)
  B/Malaysia[CD4-CD40L] D21 (N=44;36;35) | 858.29 (562.66) | 648.87 (571.71) | 748.64 (673.49)
  Pool FLU[CD4-CD40L] D0 (N=44;36;36) | 987.45 (890.57) | 923.21 (555.48) | 1625.21 (968.97)
  Pool FLU[CD4-CD40L] D0 (N=44;36;35) | 1941.32 (1283.08) | 1399.44 (1125.57) | 1891.90 (1180.76)
  A/Solomon Islands[CD4-IFNγ] D0 (N=44;36;36) | 225.18 (246.92) | 178.68 (209.78) | 321.79 (394.96)
  A/Solomon Islands[CD4-IFNγ] D21 (N=44;36;35) | 444.36 (446.32) | 297.00 (380.68) | 276.77 (478.52)
  A/Wisconsin[CD4-IFNγ] D0 (N=44;36;36) | 327.24 (327.82) | 280.71 (243.51) | 431.80 (490.54)
  A/Wisconsin[CD4-IFNγ] D21 (N=44;36;35) | 594.70 (547.10) | 425.95 (366.97) | 374.53 (618.57)
  B/Malaysia[CD4-IFNγ] D0 (N=44;35;36) | 314.05 (343.68) | 254.50 (268.96) | 471.54 (429.46)
  B/Malaysia[CD4-IFNγ] D21 (N=44;36;35) | 565.96 (386.51) | 395.62 (445.62) | 612.24 (529.06)
  Pool FLU[CD4-IFNγ] D0 (N=44;36;36) | 702.42 (642.37) | 575.66 (442.31) | 924.86 (704.75)
  Pool FLU[CD4-IFNγ] D21 (N=44;36;35) | 1231.82 (926.67) | 892.48 (794.53) | 1108.49 (956.85)
  A/Solomon Islands[CD4-IL2] D0 (N=44;36;36) | 253.44 (281.09) | 146.65 (216.35) | 314.65 (418.81)
  A/Solomon Islands[CD4-IL2] D21 (N=44;36;35) | 616.24 (527.94) | 386.68 (403.33) | 278.09 (479.01)
  A/Wisconsin[CD4-IL2] D0 (N=44;36;36) | 500.73 (465.55) | 425.33 (377.19) | 735.18 (560.20)
  A/Wisconsin[CD4-IL2] D21 (N=44;36;35) | 836.51 (650.10) | 649.78 (561.75) | 507.19 (747.26)
  B/Malaysia[CD4- IL2] D0 (N=44;35;36) | 423.52 (454.12) | 317.95 (314.42) | 598.54 (495.94)
  B/Malaysia[CD4- IL2] D21 (N=44;36;35) | 837.64 (530.27) | 609.36 (501.15) | 797.20 (619.24)
  Pool FLU[CD4-IL2] D0 (N=44;36;36) | 861.71 (826.31) | 852.92 (562.42) | 1398.63 (889.24)
  Pool FLU[CD4-IL2] D21 (N=44;36;35) | 1711.92 (1141.42) | 1253.42 (962.58) | 1643.55 (1047.94)
  A/Solomon Islands[CD4-TFNα] D0 (N=44;36;36) | 213.84 (261.37) | 157.07 (191.42) | 257.79 (414.20)
  A/Solomon Islands[CD4-TFNα] D21 (N=44;36;35) | 438.22 (458.26) | 200.94 (422.70) | 234.56 (509.44)
  A/Wisconsin[CD4-TFNα] D0 (N=44;36;36) | 505.57 (480.19) | 398.34 (330.78) | 626.76 (667.79)
  A/Wisconsin[CD4-TFNα] D21 (N=44;36;35) | 765.11 (686.36) | 567.86 (528.70) | 787.77 (804.78)
  B/Malaysia[CD4- TFNα] D0 (N=44;35;36) | 257.07 (342.41) | 180.31 (263.66) | 381.85 (435.63)
  B/Malaysia[CD4- TFNα] D21 (N=44;36;35) | 495.31 (410.07) | 304.21 (460.57) | 494.64 (550.12)
  Pool FLU[CD4-TFNα] D0 (N=44;36;36) | 700.87 (778.74) | 687.37 (473.04) | 1236.53 (885.31)
  Pool FLU[CD4-TFNα] D21 (N=44;36;35) | 1368.75 (1094.14) | 1016.67 (899.04) | 1356.89 (1093.09)

14. Secondary Outcome: The GM Number of CD8 T-cells Per Million CD8+ T-cells for Each Vaccine Strain and for Pooled Vaccine Strains Producing at Least Two Different Immune Markers or Producing Each of the Immune Markers Plus Another Immune Marker
Description: The vaccine strains included A/Solomon Islands, A/Wisconsin, B/Malaysia and Pool FLU antigens and the markers assessed were CD8-All doubles, CD40L, IFN-γ, IL-2 and TNF-α.
Time Frame: At Days 0 and 21
Population: as for outcome 8
Measure: Geometric Mean (Standard Deviation); unit: CD8 cells/10^6 CD8+ cells
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 44 | 36 | 36
CD8 cells/10^6 CD8+ cells
  A/Solomon Islands[CD8-All doubles] D0 (N=44;36;36) | 2.26 (136.77) | 3.28 (101.08) | 4.14 (186.27)
  A/Solomon Islands[CD8-All doubles] D21 (N=44;36;35 | 1.84 (88.15) | 1.92 (55.86) | 3.60 (138.60)
  A/Wisconsin[CD8-All doubles] D0 (N=43;36;36) | 2.75 (60.50) | 5.30 (264.71) | 2.44 (39.72)
  A/Wisconsin[CD8-All doubles] D21 (N=44;36;35) | 2.04 (65.79) | 2.55 (54.17) | 3.69 (62.67)
  B/Malaysia[CD8-All doubles] D0 (N=44;35;36) | 3.28 (159.00) | 4.12 (154.66) | 2.39 (72.34)
  B/Malaysia[CD8-All doubles] D21 (N=44;36;35) | 3.03 (89.02) | 2.69 (83.37) | 2.28 (44.43)
  Pool FLU[CD8-All doubles] D0 (N=44;36;36) | 8.91 (213.18) | 10.47 (89.43) | 9.43 (153.80)
  Pool FLU[CD8-All doubles] D21 (N=44;36;35) | 9.98 (149.19) | 8.02 (158.53) | 6.50 (95.79)
  A/Solomon Islands[CD8-CD40L] D0 (N=44;36;36) | 2.17 (124.96) | 1.97 (88.18) | 1.61 (22.41)
  A/Solomon Islands[CD8-CD40L] D21 (N=44;36;35) | 1.43 (40.80) | 1.64 (30.98) | 1.94 (47.82)
  A/Wisconsin[CD8-CD40L] D0 (N=43;36;36) | 2.14 (32.90) | 2.67 (222.75) | 1.70 (35.64)
  A/Wisconsin[CD8-CD40L] D21 (N=44;36;35) | 1.52 (45.12) | 1.68 (40.13) | 2.55 (44.60)
  B/Malaysia[CD8-CD40L] D0 (N=44;35;36) | 3.44 (150.26) | 2.27 (96.08) | 2.49 (57.45)
  B/Malaysia[CD8-CD40L] D21 (N=44;36;35) | 2.49 (90.52) | 1.62 (40.21) | 2.59 (45.37)
  Pool FLU[CD8-CD40L] D0 (N=44;36;36) | 7.70 (171.70) | 6.52 (67.52) | 4.42 (49.26)
  Pool FLU[CD8-CD40L] D21 (N=44;36;35) | 4.92 (129.03) | 4.64 (135.66) | 3.41 (60.34)
  A/Solomon Islands[CD8-IFNγ] D0 (N=44;36;36) | 2.07 (36.81) | 1.49 (49.87) | 3.15 (173.10)
  A/Solomon Islands[CD8-IFNγ] D21 (N=44;36;35) | 1.77 (72.15) | 2.12 (38.86) | 3.53 (113.89)
  A/Wisconsin[CD8-IFNγ] D0 (N=43;36;36) | 1.71 (31.52) | 2.76 (45.51) | 1.27 (16.73)
  A/Wisconsin[CD8-IFNγ] D21 (N=44;36;35) | 1.80 (26.18) | 2.73 (55.42) | 1.88 (33.19)
  B/Malaysia[CD8-IFNγ] D0 (N=44;35;36) | 1.93 (47.54) | 2.75 (135.21) | 2.43 (53.85)
  B/Malaysia[CD8-IFNγ] D21 (N=44;36;35) | 2.15 (35.22) | 2.24 (59.72) | 1.47 (19.69)
  Pool FLU[CD8-IFNγ] D0 (N=44;36;36) | 2.86 (46.18) | 2.48 (50.62) | 3.88 (117.16)
  Pool FLU[CD8-IFNγ] D21 (N=44;36;35) | 2.55 (47.59) | 4.17 (75.18) | 2.57 (50.74)
  A/Solomon Islands[CD8-IL2] D0 (N=44;36;36) | 2.17 (135.16) | 3.16 (92.06) | 2.49 (125.60)
  A/Solomon Islands[CD8-IL2] D21 (N=44;36;35) | 1.54 (76.05) | 1.46 (28.82) | 4.26 (129.70)
  A/Wisconsin[CD8-IL2] D0 (N=43;36;36) | 2.55 (65.54) | 4.58 (263.11) | 1.69 (30.56)
  A/Wisconsin[CD8-IL2] D21 (N=44;36;35) | 2.30 (65.28) | 1.87 (46.74) | 2.95 (74.62)
  B/Malaysia[CD8-IL2] D0 (N=44;35;36) | 2.35 (136.20) | 3.18 (142.54) | 1.90 (32.04)
  B/Malaysia[CD8-IL2] D21 (N=44;36;35) | 3.12 (97.43) | 2.36 (73.10) | 3.69 (50.07)
  Pool FLU[CD8-IL2] D0 (N=44;36;36) | 7.71 (210.95) | 8.20 (96.31) | 6.61 (63.15)
  Pool FLU[CD8-IL2] D21 (N=44;36;35) | 9.19 (155.66) | 8.89 (149.48) | 5.36 (73.11)
  A/Solomon Islands[CD8-TFNα] D0 (N=44;36;36) | 2.42 (49.99) | 1.99 (70.11) | 3.75 (175.10)
  A/Solomon Islands[CD8-TFNα] D21 (N=44;36;35) | 1.97 (68.53) | 2.40 (41.63) | 2.99 (132.56)
  A/Wisconsin[CD8-TFNα] D0 (N=43;36;36) | 3.54 (76.40) | 5.58 (70.98) | 2.44 (44.31)
  A/Wisconsin[CD8-TFNα] D21 (N=44;36;35) | 2.84 (42.13) | 2.76 (65.68) | 2.19 (48.45)
  B/Malaysia[CD8-TFNα] D0 (N=44;35;36) | 2.73 (80.16) | 8.42 (104.25) | 2.38 (72.34)
  B/Malaysia[CD8-TFNα] D21 (N=44;36;35) | 2.76 (52.39) | 3.42 (64.32) | 1.66 (30.79)
  Pool FLU[CD8-TFNα] D0 (N=44;36;36) | 6.74 (92.88) | 8.70 (72.98) | 3.32 (142.50)
  Pool FLU[CD8-TFNα] D21 (N=44;36;35) | 5.86 (58.58) | 5.55 (104.44) | 4.56 (70.82)

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed up to day 21. Systematically assessed frequent adverse events (AEs) and Non-systematically assessed frequent AEs were assessed during 7 day and 21 day post-vaccination period respectively.
Description: For the frequent adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | Adjuvanted Influenza Vaccine GSK576389A Group | Fluarix Elderly Group | Fluarix Young Group
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 46/55 | 24/40 | 36/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adjuvanted Influenza Vaccine GSK576389A Group (N=55) | Fluarix Elderly Group (N=40) | Fluarix Young Group (N=38)
Pain (General disorders) | 40 | 12 | 34
Redness (General disorders) | 13 | 6 | 1
Swelling (General disorders) | 6 | 4 | 0
Arthralgia (General disorders) | 6 | 6 | 2
Fatigue (General disorders) | 19 | 6 | 9
Headache (General disorders) | 13 | 5 | 8
Myalgia (General disorders) | 10 | 3 | 10
Nausea (General disorders) | 4 | 0 | 3
Shivering (General disorders) | 10 | 0 | 2
Temperature (General disorders) | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Rhinitis (Infections and infestations) | 2 | 1 | 2
Gastroenteritis (Infections and infestations) | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 0 | 3
Influenza like illness (General disorders) | 0 | 0 | 3
Injection site pruritus (General disorders) | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.